CLINICAL TRIAL: NCT02005107
Title: A Comparison of Immediate and Extended Release Venlafaxine Following Bariatric Surgery
Brief Title: Venlafaxine PK Following Bariatric Surgery
Acronym: VLX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: North Dakota State University (Other)
Collaborators: Neuropsychiatric Research Institute, Fargo, North Dakota (Other)
Responsible Party: Principal Investigator, Kristine Steffen, Associate Professor, North Dakota State University, North Dakota State University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: KSteffenVLX; EPSCOR (Other: North Dakota State University)
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Roux en Y Gastric Bypass; Sleeve Gastrectomy
MeSH Terms: interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- venlafaxine (Experimental): Venlafaxine IR and XR, single dosages of each separated by a wash-out period
  Interventions: Drug: Venlafaxine IR and Venlafaxine XR
- Venlafaxine XR and Venlafaxine IR (Other): Each participant (3 groups of participants) will receive one dose of venlafaxine IR and one dose of venlafaxine XR seperated by a wash-out period.
  Interventions: Drug: Venlafaxine IR and Venlafaxine XR

INTERVENTIONS:
Drug: Venlafaxine IR and Venlafaxine XR
  Other Names: Effexor and Effexor XR

SUMMARY:
This study is being conducted to evaluate how the body absorbs and processes the immediate release (IR) and sustained release (XR) medication venlafaxine (Effexor®). Subject who are 1-3 years post gastric bypass or sleeve gastrectomy surgery will be invited to participate. Non-surgical controls will also be enrolled based on a matching criteria to post gastric bypass subjects. Participants will be asked to complete two 12-hour study days approximately 11 days apart. This study will enroll up to 30 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Age 18-65 (inclusive, at time of informed consent)
3. No tobacco use in the past three months.
4. Underwent Roux-en-Y Gastric Bypass or Sleeve Gastrectomy weight loss surgery 12-36 months prior to study OR has not had a weight loss surgery but matches the gastric bypass patients on age, gender, and BMI. Criteria for matching will be established at the beginning of the study in consultation with the statistical team and addressed as needed with the input of the biostatistician.
5. Ability to read, write and understand English

Exclusion Criteria:

1. Taking a medication that has a clinically significant interaction with venlafaxine or an interaction that may alter the study data.
2. Hypersensitivity to venlafaxine or any excipient contained within the dosage forms
3. Inability to tolerate repeated blood draws.
4. Any history of bipoloar disorder or a psychotic disorder.
5. Current major depressive disorder or current suicidality.
6. Alcohol or substance dependence in the past year.
7. Currently pregnant or lactating or unwillingness to use medically accepted contraception during study
8. Taking a medication which significantly alters gastrointesinal transit time or significantly reduces acid secretion (e.g. routine use of proton pump inhibitors, H2 antagonists, sucralfate).
9. Medical conditon which may increase participant risk with venlafaxine or uncontrolled hypertension at the discretion of the examining provider.
10. Hepatic insufficiency as defined by any hepatic enzyme greater than 3x the upper limit of normal or other hepatic laboratory abnormalities at the discretion of the medical provider.
11. Renal impairment as evidence by a calculated creatinine clearance of less than or equal to 70ml/min or other abnormality on a renal panel that the medical provider feels puts the participant at risk.
12. Poor or ultra-rapid Cytochrome P450 2D6 metabolizer.
13. Self reported history of viral hepatits or HIV.
14. Positive urine drug screen unless documented prescription of a non-interacting medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Venlafaxine Plasma Concentrations/Area-Under-the-Curve (AUC) | 24 hours intervals
  The primary aim of this research is to provide a comparison of pharmacokinetic measures associated with a single dose of venlafaxine IR (immediate release) and venlafaxine XR (sustained release) in Roux-en-Y Gastric Bypass, Sleeve Gastrectomy, and matched nonsurgical "control" subjects. Comparisons will be based upon venlafaxine plasma concentrations obtained during the 24 hour sample collection window.

SECONDARY OUTCOMES:
Secondary PK Characteristics (Composite) | 24 hour collection
  We will also evaluate other PK characteristics associated with venlafaxine, such as Cmax, Tmax, t1/2, and the ratio of venlafaxine to the active metabolite ODV, and others.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine J Steffen, Pharm.D., Ph.D., Principal Investigator — North Dakota State University & Neuropsychiatric Research Institute
Locations (1):
- Neuropsychiatric Research Institute, Fargo, North Dakota, United States

REFERENCES:
- See also: Neuropsychiatric Research Institute Website — http://www.nrifargo.com